

## İNÖNÜ UNIVERSITY HEALTH SCIENCES NON-INTERVENTIVE CLINICAL RESEARCH AND PUBLICATION ETHICS COMMITTEE INFORMATIVE CONSENT FORM



You Prof. Dr. We invite you to the research titled "The Effect of Therapeutic Touch and Music Concert on Sleep Quality, Menopausal Symptoms and Quality of Life in Menopausal Women" conducted by Fatma KESKİN under the consultancy of Yurdagül YAĞMUR. Before deciding whether or not to participate in this research, you need to know why and how the research will be conducted. Therefore, it is very important to read and understand this form. If there is something that you do not understand and is not clear to you, or if you want more information, ask us.

Participation in this study is completely voluntary. You have the right to refuse to participate in the study or to withdraw from the study at any time after participating. Participants/Volunteers under the age of 18 were informed by making necessary explanations to their legal representatives in their Custody or Guardianship. Required Permission/Consent was obtained for the study. Your participation in the study, answering the questions means that you give your consent / consent to participate in the research. Do not be under pressure or suggestion from anyone while answering the questions on the forms given to you. The information obtained from these forms will be used for research purposes only. Even if the research is published, your name and identity information will remain strictly confidential and will not be given to a third party.

Address and Telephones of your Researcher, who can be reached 24 hours a day, whenever you want: İnönü University, Faculty of Nursing, Department of Gynecology and Diseases / MALATYA

Cep: 0544 817 14 44



## İNÖNÜ UNIVERSITY HEALTH SCIENCES NON-INTERVENTIVE CLINICAL RESEARCH AND PUBLICATION ETHICS COMMITTEE INFORMATIVE CONSENT FORM



## CONSENT TO PARTICIPATE IN THE RESEARCH

I have read the information above and should be given to the participant/volunteer before the research and I fully understand the scope and purpose of the study I am asked to participate in, and my responsibilities as a volunteer. Written and verbal explanation about the study was made by the researcher whose name is mentioned below. I had the opportunity to ask questions and discuss and got satisfactory answers. To me; The possible risks and benefits of the study were also explained orally. I understood that I could leave this work whenever I wanted and without having to give any reason, and that I would not face any negative consequences if I quit.

| VOLUNTEER | SIGNATURE/DATE |
|------------------|----------------|
| NAME AND SURNAME | |
| ADDRESS | |
| Phone | |
| DATE | |

| RESEARCHER | | SIGNATURE/DATE |
|---|---|---|
| ADI-SOYADI ve GÖREVİ | Fatma KESKİN | |
| ADRES | İnönü University, Faculty of Nursing, Department of Women's Health and Diseases | |
| TELEFON | 05448171444 | |
| TARİH | | |